CLINICAL TRIAL: NCT07181486
Title: Phase 1 Randomized Double-Blind Placebo-Controlled Safety Study of MucoCept-CVN (Lactobacillus Jensenii 1153-1666) Administered Vaginally to Healthy Women
Brief Title: Safety Study of MucoCept-CVN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Craig Cohen, MD, MPH (Other)
Collaborators: Osel, Inc. (Industry); Duke University (Other); DFNet Research Inc. (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Craig Cohen, MD, MPH, Professor, Obstetrics, Gynecology, and Reproductive Sciences, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: U01AI186333 (NIH); U01AI186333 (NIH)
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: HIV -1 Infection
Keywords: HIV prevention; live biotherapeutic product; MucoCept-CVN; Vaginal microbiome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For this first-in-human study, the first two participants for single dose (Cohort 1) and triple dose (Cohort 3) are unblinded and will receive the investigational product MucoCept-CVN.
  Cohort 2 (single dose randomized) and Cohort 4 (triple dose randomized) are double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single Dose MucoCept-CVN (Active Comparator): Two women in Cohort 1 will receive a single dose of active investigational product. Two of four women in Cohort 2 (1:1 randomization) will receive a single doses of active investigational product.
  Interventions: Drug: Live Biotherapeutic Product L. jensenii 1153-1666
- Triple Dose MucoCept-CVN (Active Comparator): Two women in Cohort 3 will receive three doses of active investigational product. Two of four women in Cohort 4 (1:1 randomization) will receive three doses of active investigational product.
  Interventions: Drug: Live Biotherapeutic Product L. jensenii 1153-1666
- Placebo (Single Dose and Triple Dose) (Placebo Comparator): Two of four women in Cohort 2 (1:1 randomization) will receive one dose of placebo.
  Two of four women in Cohort 4 (1:1 randomization) will receive three dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Live Biotherapeutic Product L. jensenii 1153-1666 — The vaginally administered MucoCept-CVN contains Lactobacillus jensenii 1153-1666, a natural component of the human vaginal microbiota that has been modified to continuously express the potent HIV entry inhibitor modified-cyanovirin-N (mCV-N) right at the site of infection.
  MucoCept-CVN is supplied as a prefilled vaginal applicator containing Lactobacillus jensenii 1153-1666, a modified strain of L. jensenii 1153 by integrating a modified cyanovirin-N gene into its chromosome to enhance the strain's ability to inhibit HIV. Each applicator contains 200 mg of MucoCept-CVN powder (1 x 109 CFU), and an inactive preservation matrix.
  Arms: Single Dose MucoCept-CVN; Triple Dose MucoCept-CVN
Drug: Placebo — Each placebo applicator contains 200 mg of placebo powder comprising the same inactive ingredients of the preservation matrix as the study product.
  Arms: Placebo (Single Dose and Triple Dose)

SUMMARY:
MucoCept-CVN uses a Lactobacillus strain native to the human vagina that is modified into a live biotherapeutic product (LBP) that continuously expresses a potent anti-HIV drug. If research shows that MucoCept-CVN is safe and effective, it could become a self-renewing, female-initiated prevention product for women that promotes vaginal health and provides protection from HIV.

The goal of this first-in-human Phase 1 dose-ranging, randomized, placebo-controlled study of MucoCept-CVN is to collect data on safety, colonization, changes to the vaginal microbiota and clearance of the strain with antibiotics.

Twelve healthy women will be enrolled and take either one or three doses of MucoCept-CVN or placebo, and a week later will receive antibiotics to clear the Lactobacillus strain.

If research shows that MucoCept-CVN is safe and effective, it could become a self-renewing, long-acting, female-initiated prevention product for women that promotes vaginal health and provides protection from HIV.

DETAILED DESCRIPTION:
The goal of this first-in-human Phase 1 dose-ranging, randomized, placebo-controlled study is to collect critical data needed to advance the clinical development of MucoCept-CVN, specifically (1) understanding factors that influence vaginal colonization by L. jensenii 1153-1666, including dose and endogenous vaginal microbiota; and (2) pharmacokinetic, tissue and systemic effects of L. jensenii 1153-1666, such as adverse events (AE) and findings in colposcopy and vaginal biopsy, and (3) changes to the vaginal microbiota. We also need to show that (4) L. jensenii 1153-1666 can be sufficiently cleared with antibiotics should the need arise for rescue therapy.

Twelve healthy women will be enrolled. Two women in Cohort 1 will receive one dose of active investigational product. Four women in Cohort 2 will be randomized 1:1 to either receive one dose of active investigational product or placebo. Two women in Cohort 3 will receive three doses of active investigational product. Four women in Cohort 4 will be randomized 1:1 to either receive three doses of active investigational product or placebo. Participants will be closely followed over the course of 23-37 days until antibiotic clearance of L. jensenii 1153-1666 is achieved, with a final follow-up visit occurring 30 days after clearance (Day 53-67).

Any sexual partners of study participants will be informed and consented before enrollment of study participants, and need to agree to sexual abstinence during the study. Should exposure to L. jensenii 1153-1666 occur in sexual partners, they will receive testing for L. jensenii 1153-1666 and antibiotic clearance as safety management.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pre-menopausal women 18-45 years of age, inclusive, with regular predictable menstrual cycles
2. Ability to read and consent in English
3. Previous experience of gynecological examinations
4. Consent to participate and adhere to all procedures, including frequent visits at the UCSF Clinical Research Center (CRC) facility for at least 53 days
5. Agree to get tested for STIs and a Pap Smear
6. Agree not to use any other vaginal product during the course of the study, including spermicides
7. Agree to sexual abstinence (no vaginal, anal, and receptive oral intercourse) until the elimination of L. jensenii 1153-1666 is confirmed and for 12 hours prior to the final study visit after clearance is confirmed
8. For participants with male sexual partners: Agree to use two forms of contraception, condoms plus hormonal or permanent method (intrauterine device [IUD] or tubal ligation) during vaginal intercourse from the time clearance is established to the Final Visit 30 days after clearance. Use of spermicides is not permitted.
9. For participants with female sexual partners: Agree to use female condoms during intercourse from the time clearance is established to the Final Visit 30 days after clearance. Use of hormonal or permanent method of contraception (IUD or tubal ligation) is not required.
10. Agree to inform their sexual partner about the goals of the study and importance of sexual abstinence (no vaginal, anal, and receptive oral intercourse) and present with their partner at enrollment visit for separate consent procedure for partners

Current sexual partners of participants must meet all the following criteria to be enrolled:

1. Ability to read and consent in English
2. Consent to participate and adhere to all procedures for sexual partners should exposure to L. jensenii 1153-1666 be suspected, including multiple visits at the UCSF Clinical Research Center (CRC)
3. Agree to sexual abstinence (no vaginal, anal, and receptive oral intercourse) until the elimination of L. jensenii 1153-1666 is confirmed, and for 12 hours prior to the final study visit after clearance is confirmed

Exclusion Criteria:

1. Urogenital infection, including UTI, Trichomonas vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis, Treponema pallidum, HIV-1/2, BV, or vulvovaginal candidiasis
2. Abnormal Pap smear result
3. Pregnancy or within two months of last pregnancy or lactation
4. Antibiotic or antifungal therapy (vaginal or systemic) within 30 days of enrollment
5. Investigational or immune-suppressive drug use within 30 days of enrollment visit or 10 half-lives, or planned during the study
6. Intrauterine device insertion or removal, pelvic surgery, cervical cryotherapy, cervical laser or loop electrosurgical procedure, abortion, labioplasty within three months prior to enrollment
7. Findings during the pelvic exam at the enrollment visit involving significant deep disruption of the epithelium (e.g., Herpes genitalis lesions)
8. Known allergy to any component used in MucoCept-CVN or clindamycin and azithromycin in participant or sexual partner(s), including azithromycin-associated cholestatic jaundice.
9. History of transplant surgery, cancer, HIV, diabetes or condition that could facilitate the growth of microorganisms
10. Recent history of drug or alcohol abuse
11. Unwillingness to abstain from sexual activity during study by participant or sexual partner(s)
12. If in a sexual relationship, inability to present with their sexual partner before enrollment
13. If in a sexual relationship, having multiple concurrent partners or anonymous partners.
14. Any other condition which the study clinician feels would limit the participant's ability to be an appropriate study subject
15. History of regional enteritis (Crohn's disease), ulcerative colitis, or "antibiotic-associated" colitis

For sexual partners of study participants, the following exclusion criteria apply:

1. Known allergy to any component used in MucoCept-CVN or clindamycin and azithromycin, including azithromycin-associated cholestatic jaundice.
2. Having multiple concurrent sex partners or anonymous sex partners.
3. HIV-1/2 infection
4. Any other condition which the study clinician feels would limit the ability of sexual partner(s) to complete the study
5. Co-enrollment in clinical trials testing study drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety of MucoCept-CVN - Adverse Events | From enrollment to the end of follow up at 8 weeks
  Proportion of participants with serious adverse events, any genital AEs and Grade 2 or above systemic AEs.
Antibiotic Clearance of L.jensenii 1153-1666 | From enrollment to the end of follow up at 8 weeks
  Inability to clear L. jensenii 1153-1666 after administration of antibiotics, using next generation sequencing (NGS).

SECONDARY OUTCOMES:
Safety of MucoCept-CVN - Vaginal Inflammation | From enrollment to the end of follow up at 8 weeks
  Proportion of participants with colposcopic findings and inflammation in vaginal biopsy.
Vaginal Colonization with L. jensenii 1153-1666 | From enrollment to the end of follow up at 8 weeks
  Proportion of participants with achieved vaginal colonization and clearance of vaginal colonization with L. jensenii 1153-1666, using next generation sequencing (NGS).
Tolerability - Proportion of participants not stopping the study due to Adverse Events | From enrollment to the end of follow up at 8 weeks
  Tolerability as proportion of participants not stopping the study due to AE.
Acceptability | From enrollment to the end of follow up at 8 weeks
  Acceptability of MucoCept-CVN using a self-administered questionnaire at enrollment and final visit, including perceptions around method of delivery and dosing, and self-reported attitudes about positive and negative study product attributes.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Cohen, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing the value and further advancement of this research and we plan to make the data available as widely and freely as possible, while safeguarding the privacy of participants. Therefore, we will provide qualified researchers access to the data in a timely manner after main findings from the final dataset have been accepted for publication.
  The proposed research will include data from female subjects, including current medical history, concomitant medication information (including concurrent use of contraceptives), stage of menstrual cycle, and behavioral data (e.g. sexual behavior, douching and genital hygiene practices). In addition, there will be a comprehensive database of laboratory data, including results on strain colonization, measurement of CV-N in blood and vaginal fluid, and HIV infectivity assay results, etc.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 01 May 2028 - 30 April 2033
Access Criteria: We will provide qualified researchers access to the data after main findings from the final dataset have been accepted for publication.
  We will remove identifiers from the datasets prior to release and will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed and (4) ethical committee approval from the UCSF IRB.

REFERENCES:
- See also: study recruitment website — https://www.mucocept.com/